CLINICAL TRIAL: NCT00516711
Title: Role of Volatile Anesthetics for Hepatic Protection in Ischemia-reperfusion
Brief Title: Role of Volatile Anesthetics for Hepatic Protection
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Zurich (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: StV 5-2006
Record Dates: First submitted 2007-08-14; First posted 2007-08-15 (Estimated); Last update posted 2010-09-15 (Estimated); Status verified 2007-08

CONDITIONS: Reperfusion Injury
Keywords: Surgery with Pringle maneuver needed for liver resection
MeSH Terms: conditions — Reperfusion Injury | interventions — Sevoflurane

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Sevoflurane

SUMMARY:
This study aims to evaluate the attenuation of ischemic-reperfusion injury in the liver after sevoflurane preconditioning. In the presence of sevoflurane, an attenuation of liver injury is hypothesized (diminished increase of liver enzymes, reduced production of inflammatory mediators).

DETAILED DESCRIPTION:
Organ protection; preconditioning; volatile anesthetics; ischemia reperfusion

ELIGIBILITY:
Inclusion Criteria:

* Older than 18 years of age
* Patients undergoing liver resection (benign or malignant tumors)

Exclusion Criteria:

* Laparoscopic liver resection coagulopathy (platelets < 50,000/ml, Quick < 50%)
* Liver cirrhosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Dates: Start 2006-03; Primary Completion 2007-12 (Actual); Study Completion 2007-12 (Actual)

PRIMARY OUTCOMES:
Blood levels of aspartate aminotransferase (AST), alanine aminotransferase (ALT)

CONTACTS AND LOCATIONS:
Overall Officials: 01 Studienregister MasterAdmins, Study Director — UniversitaetsSpital Zuerich
Locations (1):
- University Hospital of Zurich, Zurich, Switzerland

REFERENCES:
- [Derived] Beck-Schimmer B, Breitenstein S, Urech S, De Conno E, Wittlinger M, Puhan M, Jochum W, Spahn DR, Graf R, Clavien PA. A randomized controlled trial on pharmacological preconditioning in liver surgery using a volatile anesthetic. Ann Surg. 2008 Dec;248(6):909-18. doi: 10.1097/SLA.0b013e31818f3dda. PMID 19092335